CLINICAL TRIAL: NCT07156396
Title: Comparative Evaluation of A Novel Anesthetic Device vs. Conventional Infiltration in Pain Perception Among A Group of Pediatric Patients Undergoing Extraction Of Mandibular Primary Molars: A Randomized Clinical Trial
Brief Title: SleeperOne vs. Conventional Infiltration: Pain Perception in Mandibular Primary Molar Extraction
Acronym: SOTIMAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ameera Alaa Eldin Abdalazim Khalifa (Other)
Responsible Party: Sponsor-Investigator, Ameera Alaa Eldin Abdalazim Khalifa, MSc Candidate in Pediatric Dentistry, Faculty of Dentistry, Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 832025
Record Dates: First submitted 2025-08-08; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-07

CONDITIONS: Dental Anxiety; Pain; Pain Management; Extraction, Tooth
Keywords: Pediatric dentistry; Tooth extraction; conventional infiltration; sleeperOne 5; Computer-Controlled anesthesia; Pain Perception
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Infiltration (Active Comparator): Children will receive 3% mepivacaine with conventional syringe after 20% benzocaine
  Interventions: Procedure: Conventional Infiltration
- SleeperOne® Device (Experimental): Children will receive 3% mepivacaine using SleeperOne® device after 20% benzocaine.
  Interventions: Device: SleeperOne®, dental Hitec, France

INTERVENTIONS:
Device: SleeperOne®, dental Hitec, France — SleeperOne® is a computerized local anesthetic delivery system used to deliver 3% mepivacaine following application of 20% benzocaine topical gel. It is designed to reduce injection pain and improve comfort during pediatric dental procedures.
  Arms: SleeperOne® Device
Procedure: Conventional Infiltration — Local anesthetic (3% mepivacaine) will be administered using a conventional dental syringe after the application of 20% benzocaine topical anesthetic.
  Arms: Conventional Infiltration

SUMMARY:
This clinical trial is being conducted in the Department of Pediatric Dentistry, Faculty of Dentistry, Cairo University. The purpose of the study is to compare the pain perception and comfort of children during tooth extraction when using a computer-controlled local anesthetic device (SleeperOne® 5) versus the conventional syringe infiltration technique.

Children between 3 and 5 years of age who require extraction of a maxillary primary molar will be invited to participate. Before starting, a topical anesthetic gel (benzocaine) will be applied. Then, local anesthesia will be given using either the SleeperOne® device or the traditional syringe, depending on the group assigned.

Pain during injection and extraction will be assessed using both child-friendly rating scales and independent evaluation by the dentist. Patient anxiety, heart rate, and blood pressure will also be recorded.

This study aims to provide evidence on whether computer-controlled anesthesia can reduce children's pain and anxiety compared with the conventional method, leading to a more comfortable dental experience.

The study is a randomized clinical trial and will be conducted in a single visit at the Pediatric Dentistry Outpatient Clinic, Faculty of Dentistry, Cairo University. The results may help improve pain management and patient comfort during dental treatment for children.

DETAILED DESCRIPTION:
This randomized clinical trial aims to evaluate and compare the pain perception and anxiety levels associated with the use of a computer-controlled local anesthetic delivery system (SleeperOne®) versus conventional local infiltration using a standard syringe in pediatric patients undergoing extraction of mandibular primary molars.

A total of 28 healthy children aged 3 to 5 years, requiring extraction of at least one mandibular primary molar, will be enrolled and randomly assigned into two parallel groups: the intervention group (SleeperOne®) and the control group (conventional syringe). Both groups will receive the same anesthetic solution: 3% Mepivacaine without vasoconstrictor. Topical anesthesia will be applied using 20% benzocaine gel before injection in all participants.

Pain management during dental treatment in children is a major concern in pediatric dentistry. Traditional infiltration anesthesia using a syringe is effective but often associated with pain, anxiety, and fear, which can negatively affect child cooperation. Computer-controlled local anesthetic delivery (CCLAD) systems, such as the SleeperOne® 5, have been developed to minimize these issues by providing a slow and steady flow of anesthesia with improved ergonomics for the operator.

This randomized clinical trial will compare pain perception during maxillary primary molar extraction in children using the SleeperOne® 5 device versus conventional infiltration with a standard dental syringe. The trial will follow a parallel design with two arms: an intervention group receiving local anesthesia via the SleeperOne® 5, and a control group receiving conventional syringe infiltration.

Participants will be children aged 3-5 years who require extraction of a maxillary primary molar. Topical anesthesia with benzocaine will be applied prior to injection in both groups. Local infiltration will then be administered using either the SleeperOne® 5 or a conventional syringe, depending on group allocation.

The primary outcome is pain perception during injection and extraction, measured subjectively using the Wong-Baker Faces Pain Rating Scale (WBFPRS) and objectively using the Sound, Eye, and Motor (SEM) scale by an independent, blinded evaluator. Secondary outcomes include patient anxiety, recorded using the Modified Child Dental Anxiety Scale (MCDAS), and physiological responses (heart rate and blood pressure) measured with a digital monitor.

The study is designed with two parallel groups, with an anticipated sample size of 28 children (14 per group), based on a power calculation. Randomization will be performed using a computer-generated list. Blinding of participants is not possible due to the nature of the interventions, but outcome assessment will be blinded.

The results of this study are expected to provide clinical evidence on whether CCLAD (SleeperOne® 5) offers a significant advantage over conventional infiltration in reducing pain and anxiety during pediatric dental extractions.

ELIGIBILITY:
Inclusion criteria:

* Children Aged between 3 to 5 years.
* Medically fit children classified as ASA physical status I and II
* Parents acceptance to participate in the study (informed consent)
* Children with teeth diagnostically confirmed to require extraction

Exclusion criteria:

* Patients with an allergy to local anesthesia.
* Uncooperative children
* Children requiring general anesthesia

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2025-09-02 (Estimated); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
Pain during injection | immediately during local anesthetic injection
  Pain during injection will be assessed using the Sound-Eye-Motor (SEM) pain scale, which is a validated observational scale for evaluating pain response in pediatric patients. The SEM scale consists of three components-sound, eye, and motor reaction-each scored from 1 to 4, where a lower score indicates minimal or no pain and a higher score indicates greater discomfort. The total score is interpreted to reflect the child's behavioral reaction to the injection stimulus.

SECONDARY OUTCOMES:
Patient anxiety | During injection and extraction in the same clinical visit
  Patient anxiety will be assessed during the dental anesthesia procedure using the Modified Child Dental Anxiety Scale (MCDAS). The scale provides a subjective measure of the child's level of anxiety, scored from 8 to 40, with higher scores indicating greater anxiety.
Heart rate changes | within 15 minutes after injection
  Heart rate will be monitored using a digital pulse oximeter as an objective measure of patient anxiety. Baseline and intraoperative readings will be compared between groups.
Blood pressure changes | within 15 minutes after injection
  Blood pressure will be recorded using a digital sphygmomanometer to evaluate physiological responses to local anesthesia. Baseline and intraoperative readings will be compared.
Soft tissue injury | Within 24 hours after the procedure.
  Soft tissue injury (lip or cheek biting, trauma due to numbness) will be reported by parents/patients during follow-up. Any incidence will be documented and compared between groups.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a student-initiated academic trial, and data confidentiality will be maintained in accordance with ethical standards.

REFERENCES:
- See also: it introduces the sleeper one 5 anesthetic device — https://www.dentalhitec.com/
- Available data/document: Informed Consent Form: SleeperOne2025 — https://clinicaltrials.gov/study-protocol-pending — Study protocol will be uploaded and publicly accessible upon final approval.